CLINICAL TRIAL: NCT01366872
Title: Agility LP Ankle Arthroplasty: Clinical and Radiographic Outcomes
Brief Title: Agility LP Ankle Arthroplasty Outcomes
Status: Completed | Type: Observational
Sponsor: Orthopaedic Associates of Michigan, PC (Other)
Responsible Party: Principal Investigator, John G. Anderson, MD, Principal Investigator, Orthopaedic Associates of Michigan, PC
Other Study IDs: OAM-LP-2010
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-11

CONDITIONS: Rheumatoid Arthritis of Ankle; Osteoarthritis of Ankle; Traumatic Arthritis of Ankle
Keywords: ankle; arthritis; total ankle arthroplasty; Agility LP,
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a research study which is being done to determine the outcomes following Agility LP ankle replacement. This implant was approved by the FDA in 2007 and has been used since then with good early results. You are being asked to volunteer for this study because you have undergone Total Ankle Arthroplasty with Agility LP prosthesis. The purpose of the study is to compare the range of motion, level of pain and function during daily living prior to and after your ankle surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Can comprehend and sign the informed consent
* Patient must have undergone Agility LP ankle replacement between January 2006 to June 2008

Exclusion Criteria:

* Patient has had following procedures on the study limb within two years of TAA
* Revision of TAA
* Ankle arthrodesis
* Amputation
* Agility LP arthroplasty was done as a revision procedure for a failed TAA or as a takedown of ankle fusion.
* Any condition that, in the opinion of the investigator, makes the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male subjects over the age of 18 at the time of procedure who have undergone ankle joint replacement using the DePuy Agility LP Device.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John G Anderson, MD, Principal Investigator — Orthopaedic Associates of Michigan, PC
Locations (1):
- Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Orthopaedic clinical, Agility LP TAA
Pre-assignment Details: Minimum of 2 years post index procedure
Groups:
- Agility LP Total Ankle Arthroplasty: Patients who underwent Total Ankle Arthroplasty using the Agility LP device a minimum of 2 years prior to study enrollment.
Period: Overall Study
Arm/Group | Agility LP Total Ankle Arthroplasty
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Agility LP Total Ankle Arthroplasty
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (4.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Functional Outcomes Following Agility LP Ankle Replacement
Description: Range of Motion - Combined total of dorsiflexion and plantarflexion. Full range of motion is described as 30 degrees or more. Partial limitation is described as 29 to 15 degrees. Range of motion that is less than 15 degrees is described as severely limited.
Time Frame: A Minimum of 2 Years Post Index Procedure
Population: Per surgical history (protocol).
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Agility LP Total Ankle Arthroplasty
Number analyzed (Participants) | 50
Degrees
  Pre-operative range of motion | 37.67 (2.516)
  Post-operative range of motion | 37.07 (2.511)

2. Secondary Outcome: Evaluation of Complication and Reoperation Rates
Description: Number of reported complications/reoperations following the index procedure.
Time Frame: A Minimum of 2 Years Post Index Procedure
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | Agility LP Total Ankle Arthroplasty
Number analyzed (Participants) | 50
participants
  Hardware Complication/Removal | 6
  Wound Complication | 5
  Revisions and Takedowns | 3
  Other Surgical Intervention Related | 10
  Other Surgical Intervention Not Related | 3

3. Secondary Outcome: Radiographic Predictors of Implant Failures and Poor Outcomes
Description: Post-Operative radiographic disposition. Subsidence is described as the component sinking into the bone. Ingrowth is described as the implant components to conform into the tibia and talus.
Time Frame: A Minimum of 2 Years Post Index Procedure
Population: Per protocol, patients who were completely revised were excluded.
Measure: Number; unit: participants
Arm/Group | Agility LP Total Ankle Arthroplasty
Number analyzed (Participants) | 48
participants
  Talar Subsidence | 10
  Tibial Subsidence | 1
  Talar & Tibial Subsidence | 5
  Ingrowth of Both Components | 32

ADVERSE EVENTS:
Time Frame: Minimum of 2 years post index procedure
Description: Self reported by patient, medical record review
Arm/Group | Agility LP Total Ankle Arthroplasty
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 14/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Agility LP Total Ankle Arthroplasty (N=50)
Hardware Complication (Musculoskeletal and connective tissue disorders) | 6 (6) — Painful hardware which required post-surgical removal
Wound Complication (Infections and infestations) | 10 (10) — Patient who required wound care beyond the accepted standard of care for resolution.
Surgical Revision of Implant (Musculoskeletal and connective tissue disorders) | 3 (3) — Patients who had their initial implant revised or removed.
Other Surgical Intervention Related to Index Procedure (Musculoskeletal and connective tissue disorders) | 10 (10) — Patient required surgical intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No